CLINICAL TRIAL: NCT04955756
Title: Early Identification and Severity Prediction of Acute Respiratory Infectious Disease
Acronym: ESAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, chairman of the infectious disease department, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ESAR
Record Dates: First submitted 2021-06-18; First posted 2021-07-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Acute Respiratory Infection; Severe Pneumonia; Next Generation Sequencing; Multiplex PCR
Keywords: mNGS; Multiplex PCR; Acute Respiratory Infectious Disease; Severe Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mNGS group (Experimental)
  Interventions: Diagnostic Test: mNGS
- PCR group (Experimental)
  Interventions: Diagnostic Test: Multiplex PCR

INTERVENTIONS:
Diagnostic Test: mNGS — Participants will be randomized to receive mNGS or multiplex PCR for diagnosis at enrollment.
  Arms: mNGS group
Diagnostic Test: Multiplex PCR — Participants will be randomized to receive mNGS or multiplex PCR for diagnosis at enrollment.
  Arms: PCR group

SUMMARY:
Early identification and Severity prediction of Acute Respiratory infectious disease has become a top priority for clinicians at department of infectious and respiratory diseases after COVID-19 broke out. This is a multicenter, prospective, and randomized study, which aims to figure out the best way of early identification and severity prediction of acute respiratory infectious diseases. Patients with suspected acute respiratory infectious diseases will be enrolled into this study and received two different diagnostic pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 80 years old
2. No limits in gender
3. Patients who are newly present with cough, sputum, or exacerbated with pyogenic sputum, with or without chest pain within 2 weeks;
4. Patients who meet at least one of the following 4 requirements:

   1. fever;
   2. Sign of pulmonary consolidation or wet wales
   3. WBC>10×10^9/L or <4×10^9/L;
   4. patchy, infiltrating shadows or interstitial changes, with or without pleural effusion on chest radiological examination.

Exclusion Criteria:

1. Highly suspected or diagnosed pulmonary non-infectious disease (Tumor, Immune disease, etc.) without evidence for infection;
2. Pathogen has been identified without evidence for co-infection;
3. Insufficiency of respiratory and blood samples;
4. Patients who are unable to collaborate due to physical or mental disorders;
5. Patients who have been engaged to other clinical trials;
6. Any conditions make it unsafe for the subject to participate;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-04-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
time for targetted antibiotic treatment | 28 days
  time interval from enrollment to targetted antibiotic treatment initiation

SECONDARY OUTCOMES:
Incidence for clinical key events | 28 days
  Incidence for clinical events including tracheal intubation, tracheotomy, ECMO, and CRRT.
Incidence for clinical remission | 28 days
  Incidence for clinical remission, which achieve the following conditions for over 24 hours: ① heart rate <100bpm; ② SBP> 90mmHg; ③Body Temperature <38℃; ④ SaO2 > 90% at room temperature;
Length of hospitalization; | 28 days
  time interval between admission to hispital and discharge from the hospital when a participant is recovered
Length of ICU admission | 28 days
  time interval from admission to ICU and discharge from ICU
Length from admission to clinical events | 28 days
  time interval from admission to hospital to clinical events including tracheal intubation, tracheotomy, ECMO, and CRRT.
Sampling to Diagnosis Interval | 28 days
  time interval from Sampling to Diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, Prof, Study Chair — Department of Infectious disease, Huashan Hospital, Fudan University
Locations (3):
- China (3):
  - Central Hospital of Jingan District, Shanghai, Shanghai Municipality
  - Department of Infectious Disease, Huashan Hospital, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan G, Wang H, Zhao Y, Mao E, Li M, Wang R, Zhou F, Jin S, Zhang Z, Xu K, Xu J, Liang S, Li X, Jiang L, Zhang L, Song J, Yang T, Guo J, Zhang H, Zhou Y, Wang S, Qiu C, Jiang N, Ai J, Wu J, Zhang W. Early identification and severity prediction of acute respiratory infection (ESAR): a study protocol for a randomized controlled trial. BMC Infect Dis. 2022 Jul 20;22(1):632. doi: 10.1186/s12879-022-07552-7. PMID 35858876